CLINICAL TRIAL: NCT02644018
Title: Double Blind Randomized Placebo-controlled Multicenter Study to Evaluate Clinical Efficacy and Safety of Ingavirin®, Capsules 30 mg, in 3-6 Years Old Patients With Influenza and Other Acute Respiratory Viral Infections in the Course of Standard Therapy
Brief Title: Efficacy and Safety Study of Ingavirin® to Treat Influenza and Other Acute Respiratory Viral Infections in Patients 3-6 y.o.
Acronym: ACCORD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Collaborators: Atlant Clinical Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ING-03-02-2015
Record Dates: First submitted 2015-12-22; First posted 2015-12-31 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-02

CONDITIONS: Common Cold; Influenza
Keywords: Ingavirin; Common Cold; Influenza; Acute Respiratory Viral Infections; pediatric clinical trial; Imidazolyl ethanamide pentandioic acid
MeSH Terms: conditions — Common Cold; Influenza, Human | interventions — pentanedioic acid imidazolyl ethanamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ingavirin (Experimental): Ingavirin (Imidazolyl ethanamide pentandioic acid), capsules 30 mg daily for 5 days. The contents of one capsule of Ingavirin, capsules 30 mg should be dissolved in 50-70 ml of water at room temperature or apple juice at room temperature with mandatory stirring for 20 seconds and administered orally 1 time a day regardless of the meal.
  Interventions: Drug: Imidazolyl ethanamide pentandioic acid
- Placebo (Placebo Comparator): Placebo, capsules daily for 5 days. The contents of one capsule of placebo should be dissolved in 50-70 ml of water at room temperature or apple juice at room temperature with mandatory stirring for 20 seconds and administered orally 1 time a day regardless of the meal.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Imidazolyl ethanamide pentandioic acid
  Other Names: Ingavirin
  Arms: Ingavirin
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Ingavirin ® dosed 30 mg daily is effective and safe in the treatment of influenza and other acute respiratory viral infections in the course of standard therapy in 3-6 years old patients.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent form signed by the patient's parent/adoptive parent to participate in the clinical study.
* Male and female patients aged 3-6.
* Patients with moderate course of influenza or other acute respiratory viral infections.
* Patients with clinically diagnosed influenza or other ARVI based on the body temperature > 37,5 ° C, not less than 1 of the following other symptoms of intoxication and not less than 1 of the following of catarrhal symptoms:

  * Intoxication symptoms: headache, malaise, myalgia, pain in the eyeballs;
  * Catarrhal symptoms: sore throat, rhinorrhea, cough, nasal congestion.
* Established diagnosis J06.9, J10, J11, in accordance with ICD-10.
* Uncomplicated course of influenza and other ARVI.
* Interval between onset of symptoms and enrollment to the study of not more than 36 hours.

Exclusion Criteria:

* Complicated course of influenza and other acute respiratory viral infections.
* Treatment with antiviral drugs (antivirals, interferons and interferon inducers), drugs with immunomodulatory effects or antibiotics with systemic and local action within 14 days prior to the screening visit.
* Severe influenza or other ARVI with symptoms of cardiovascular disease, and other symptoms of infectious-toxic shock, and meningoencephalitic syndromes.
* Signs of primary viral pneumonia development (presence of two or more of the following symptoms): shortness of breath, chest pain when coughing, systemic cyanosis, dullness of percussion sound at symmetrical assessment of the upper and lower parts of the lungs.
* Infectious diseases within the last week prior to enrollment.
* "RRI children" (incidence of ARVI within the last 12 months is 6 times or more).
* Asthma history.
* History of increased seizure activity.
* Severe decompensated or unstable medical or psychiatric conditions (any diseases or conditions that threaten the life of the patient or worsen the patient's prognosis and also make it impossible to conduct a clinical study in the patient).
* Cancer, HIV infection, tuberculosis, including those in history.
* Hypersensitivity to imidazolyl ethanamide pentandioic acid and/or excipients of Ingavirin product.
* Diabetes, lactose intolerance, lactase deficiency, glucose-galactose malabsorption, deficiency of sucrase/isomaltase, fructose intolerance, hereditary glucose malabsorption, deficiency of glucose-6-phosphate dehydrogenase.
* Participation of the patient in any other clinical trial within the last 90 days prior to enrollment.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 190 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Time to decrease in the Influenza and Other ARVI Severity Scale score to 2 points with no more than 1 point at individual subscales and normalization of body temperature | 5 days
  Temperature normalization means establishment of body temperature below 37 ° C without raising thereafter till 5 days after the treatment start.

SECONDARY OUTCOMES:
Time to decrease in the Influenza and Other ARVI Severity Scale score to 0 points | 5 days
Average score at the Influenza and Other ARVI Severity Scale by the 1st, 2nd, 3rd, 4th and 5th days after the start of treatment | Within 6 days from the start of treatment
The area under the "Influenza and Other ARVI Severity Scale score - time" curve by the 5th day after the start of treatment | 5 days
Time to normalization of body temperature from the start of treatment, measured in hours | 5 days
  Temperature normalization means establishment of body temperature below 37°C without raising thereafter till 5 days after the treatment start
The average body temperature by the1st, 2nd, 3rd, 4th and 5th days after the start of treatment | 5 days
The percentage of patients with normalization of body temperature by the 1st, 2nd, 3rd, 4th and 5th days after the start of treatment | 5 days
The area under the "temperature-time" curve by the 5th day after the start of treatment | 5 days
The percentage of patients with complications of influenza and other ARVI developed over the period from the 1st to the 6th and from the 1st to 14th day after the start of treatment | 14 days
The percentage of patients with severe complications of influenza and other ARVI that have developed over the period from the 1st to the 6th and from the 1st to 14th day after the start of treatment | 14 days
Time to onset of complications of influenza and other ARVI from the start of treatment | 14 days
Assessment of adverse events (AEs) and serious adverse events (SAEs) | 14 days
  Assessment of adverse events (AEs) and serious adverse events (SAEs) by means of -
  * Portion of patients who developed one or more SAE during the study
  * Portion of patients who developed one or more AE during the study
  * Portion of patients who developed one or more severe AE during the study
  * Portion of patients who developed one or more AE with definite relationship to the investigational product/ placebo during the study
  * Portion of patients who developed one or more AE with definite or probable relationship to the investigational product/ placebo during the study

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Zakharova, MD, PhD, Study Director — Valenta Pharm JSC; Yuriy V. Lobzin, MD, PhD, Principal Investigator — Scientific Research Institute of Children's Infections, Federal Biomedical Agency, Saint-Petersburg, Russian Federation
Locations (13):
- Russia (13):
  - GBOU VPO "Kazan State Medical University" of Ministry of Health of Russian Federation, Kazan'
  - GBOU VPO "Krasnoyarsk State Medical University n.a.n V.F. Voyno-Yasenetskogo" of Ministry of Health of Russian Federation, Krasnoyarsk
  - FGBU "Scientific center of children health" of the Ministry of Health of Russian Federation, Moscow
  - I.M. Sechenov First Moscow State Medical University, Moscow
  - Moscow Budgetary Public Health Facility "Infectious clinical hospital #1" of Moscow City Health Department, Moscow
  - GBOU VPO "Novosibirsk State Medical University of Ministry of Health of Russian Federation", Novosibirsk
  - Children's city outpatients clinic № 5, Perm
  - Children's city outpatients clinic № 4, Rostov-on-Don
  - GBOU VPO "Rostov State Medical University" of Ministry of Health of Russian Federation, Rostov-on-Don
  - FGBU "Scientific Research Institute of Children's Infections, Federal Biomedical Agency", Saint Petersburg
  - FGBOU VPO "Mordov State University n.a. N.P. Ogarev", Saransk
  - GBOU VPO "Siberia State Medcial University" of Ministry of Health of Russian Federation, Tomsk
  - GBOU VPO "Yaroslavl State Medical University" of Ministry of Health of Russian Federation, Yaroslavl

IPD SHARING:
Plan to Share IPD: No